CLINICAL TRIAL: NCT03104088
Title: Studying Cognition in SPG4 Compared to Healthy Controls
Brief Title: Studying Cognition in SPG4
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ludger Schöls, Prinicipal Investigator, University Hospital Tuebingen
Other Study IDs: Cognition_SPG4
Record Dates: First submitted 2017-03-23; First posted 2017-04-07 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Cognitive Impairment; Hereditary Spastic Paraplegia
MeSH Terms: conditions — Cognitive Dysfunction; Spastic Paraplegia, Hereditary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SPG4 patients
  Interventions: Diagnostic Test: CANTAB; Diagnostic Test: MOCA
- Healthy controls
  Interventions: Diagnostic Test: CANTAB; Diagnostic Test: MOCA

INTERVENTIONS:
Diagnostic Test: CANTAB — CANTAB Cognitive Assessment (tablet based cognitive testing from CAMCOG)
Diagnostic Test: MOCA — Montreal cognitive assessment (MOCA) in German

SUMMARY:
Comparing the cognitive levels of patients with SPG4 mutations to healthy controls.

DETAILED DESCRIPTION:
Comparing the cognitive levels of patients with SPG4 mutations to healthy controls by using the CANTAB® and MoCA.

ELIGIBILITY:
Inclusion Criteria:

* Patient with SPG4 with known SPAST-Mutation (patient group) or healthy control
* Age 18 to 70 years
* Written, informed consent

Exclusion Criteria:

* Lack of ability for a written, informed consent
* Presence of gait disorder or other neurological condition (for healthy controls)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Probands will be recruited at the HSP Outpatient Clinic of the Department of Neurology in Tübingen. Eligible participants are age 18 to 70 years of age. Group 1 include p: patients with genetically confirmed SPG4 (group 1) and manifest disease with spastic gait disorder. Group 2 includes age- and sex-matched and healthy controls (spouses, other relatives or further healthy controls) with an educational level comparable to group 1 (group 2).
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-12-24 (Actual); Study Completion 2017-12-24 (Actual)

PRIMARY OUTCOMES:
Identifying cognitive affected domains by using CANTAB | day 1
  Number of SPG4 patients with affections in the examined cognitive domains by using CANTAB

CONTACTS AND LOCATIONS:
Overall Officials: Ludger Schöls, Prof. Dr., Principal Investigator — University Hospital Tübingen, Center for Neurology
Locations (1):
- University Hospital Tübingen, Center for Neurology, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rattay TW, Boldt A, Volker M, Wiethoff S, Hengel H, Schule R, Schols L. Non-motor symptoms are relevant and possibly treatable in hereditary spastic paraplegia type 4 (SPG4). J Neurol. 2020 Feb;267(2):369-379. doi: 10.1007/s00415-019-09573-w. Epub 2019 Oct 23. PMID 31646384
- See also: Article Link (DOI) — https://doi.org/10.1007/s00415-019-09573-w